CLINICAL TRIAL: NCT04280120
Title: Effect of Neural Mobilization in Bells Palsy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Lecturer, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MU-1441-99
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Bell Palsy
MeSH Terms: conditions — Bell Palsy | interventions — Massage; Exercise

STUDY DESIGN:
Intervention Model Description: The study will include a minimum of 60 participants visiting the investigator's outpatient department from 2020-2021. The equal allocation procedure will be used based on the admission of the cases.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care provider, investigator and outcome assessor will be unaware about the allocation. The therapist performing the initial assessment and the final assessment will be same but will be unaware about the patient assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Mobilisation Group (Experimental): 1. Massage therapy.
  2. Faradic electrical stimulation.
  3. Exercises in front of the mirror.
  4. Neural mobilization was applied by gently holding the lower part of the ear between the index finger and thumb. The thumb was placed at the opening of the external auditory meatus and the index finger placed behind the auricle of the ear (Figure 2). The intensity of auricular traction was determined by the patient reporting the level of discomfort. The patient tolerated 3-4 sets of gentle horizontal traction and circular movement 25 times each with 5 seconds rest.
  Interventions: Other: Neural Mobilisation; Other: Massage therapy; Diagnostic Test: Faradic electrical stimulation; Other: Exercises
- Conservative group (Active Comparator): 1. Massage therapy consisting of tapping, effleurage and finger and thumb kneading for 15-16 minutes.
  2. Faradic electrical stimulation with anode electrode at the back of the neck and cathode over the nerve trunk anterior to the earlobe. The cathodic pen electrode was used to locate the facial nerve trunk for stimulation manually. (Biphasic current, pulse time 300 microseconds, frequency 60 Hz, 20 contractions, Rest 10 seconds). The total treatment time was 15 minutes.
  3. Exercises in front of the mirror like raising the eyebrow, clinching the teeth (patient trying to see his clenched teeth in the mirror), smiling and performing other facial expressions for 12-15 minutes.
  Interventions: Other: Massage therapy; Diagnostic Test: Faradic electrical stimulation; Other: Exercises

INTERVENTIONS:
Other: Neural Mobilisation — Neural mobilization was applied by gently holding the lower part of the ear between the index finger and thumb. The thumb was placed at the opening of the external auditory meatus and the index finger placed behind the auricle of the ear (Figure 2). The intensity of auricular traction was determined by the patient reporting the level of discomfort. The patient tolerated 3-4 sets of gentle horizontal traction and circular movement 25 times each with 5 seconds rest.
  Arms: Neural Mobilisation Group
Other: Massage therapy — Massage therapy consisting of tapping, effleurage and finger and thumb kneading for 15-16 minutes.
Diagnostic Test: Faradic electrical stimulation — Faradic electrical stimulation with anode electrode at the back of the neck and cathode over the nerve trunk anterior to the earlobe. The cathodic pen electrode was used to locate the facial nerve trunk for stimulation manually. (Biphasic current, pulse time 300 microseconds, frequency 60 Hz, 20 contractions, Rest 10 seconds). The total treatment time was 15 minutes.
Other: Exercises — Exercises in front of the mirror like raising the eyebrow, clinching the teeth (patient trying to see his clenched teeth in the mirror), smiling and performing other facial expressions for 12-15 minutes.

SUMMARY:
Bells palsy is a sudden paralysis of half of the facial muscle. The BP is idiopathic and 70% responds well with drug therapy. There are many complementary therapies such as , tapping, electrical stimulation, and massage that adds to the recovery of condition. However, efficacy of neural mobilization in BP is not reported in the scientific literature.

DETAILED DESCRIPTION:
Bells Palsy responds well with drug therapy such as prednisolone and antiviral drugs for the duration of 10-12 days. However, the administration of these drugs produce adverse side effect. Therapist use a number of techniques to maintain the physiological properties of facial muscles. However, adding a new technique would add to the arsenal of techniques available for the therapist. The research is intended to determine the effect of adding Neural mobilization in the recovery of Bells Palsy. A randomized controlled trail is intended to include 60 participants divided into two groups. Experimental group will receive Neural Mobilization with conservative treatment and control group will receive conservative treatment only.

ELIGIBILITY:
Inclusion Criteria:

* The first episode of Bell's palsy.
* Modified House-Brackmann scale III-IV.

Exclusion Criteria:

* Diabetic
* Recurrent Bells palsy
* facial palsy
* History of stroke
* Any cerebrovascular accident
* epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Sunnybrook facial assessment scale | 1 year
  Sunnybrook facial assessment scale is a scale to assess quantitatively the facial asymmetry. It is a weighted scale based on evaluation of 3 different sub-scale including resting symmetry, the symmetry of voluntary movement, and severity of synkinesis to form one single composite score from 0 to 100. Firstly, the physiotherapist assesses the symmetry of the eye (0-1), cheek (0-2), and mouth (0-1) at rest. (0=normal, the weighted factor of 5). Secondly, the Physiotherapist rates facial movements during 5 standard facial expressions: a brow lift, gentile eye closure, open mouth smile, snarl and lip pucker, on a scale of 1 to 5 (1=no movement, to 5=normal movement). The values are added together and multiplied by 4. In the 3rd step, the severity of synkinesis on a 3-point scale (0=none, to 3=severe) during the 5 expressions as in the 2nd step. The overall score is given by the symmetry value of the voluntary movements minus the resting symmetry and the synkinesis.
Kinovea© tool for facial movement analysis | 1 year
  As a secondary outcome, we used Kinovea©, a free and open-source tool for movement analysis (Kinovea©, 0.8.15 2006 to 2011; Joan Charmant & Contrib, Bordeaux, France). From plain video-recordings of movements, the software allows measuring distances and times, manually or using semi-automated tracking to follow points and check live values or trajectories. Facial distances were measured after maximal contractions movements of 3 selected facial muscles: frontalis, orbicularis oris, zygomatic. A symmetry ratio calculated comparing sides of each movement pattern. Subjects had to look straight ahead towards a specified target fixed on the facing wall and it was asked them not to move during video acquisitions. It was asked to keep the head lean the wall, keeping firm it during the 3 tested movements.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - IAMR, Ghaziabad, Uttar Pradesh
  - Faizan Kashoo, Meerut, Uttar Pradesh